CLINICAL TRIAL: NCT03049059
Title: A Comparative Study for Efficacy and Safety Between 4% Hydroquinone Cream With or Without Fractional Picosecond 1,064 nm Laser for the Treatment of Dermal or Mixed Type Melasma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mae Fah Luang University Hospital (Other)
Responsible Party: Principal Investigator, Thep Chalermchai, Dr., Mae Fah Luang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 087/2559
Record Dates: First submitted 2017-02-03; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Picoseconds Laser; Melasma
MeSH Terms: conditions — Melanosis | interventions — Lasers

STUDY DESIGN:
Intervention Model Description: Randomized split face
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fractional Picosecond 1,064 nm laser and 4% hydroquinone cream (Experimental)
  Interventions: Device: Fractional Picosecond 1,064 nm laser; Drug: 4% hydroquinone cream
- 4% hydroquinone cream alone (Active Comparator)
  Interventions: Drug: 4% hydroquinone cream

INTERVENTIONS:
Device: Fractional Picosecond 1,064 nm laser — Fractional Picosecond 1,064 nm laser and daily application with 4% hydroquinone cream
  Arms: Fractional Picosecond 1,064 nm laser and 4% hydroquinone cream
Drug: 4% hydroquinone cream

SUMMARY:
A Comparative study for Efficacy and Safety Between 4% hydroquinone cream with or without Fractional Picosecond 1,064 nm Laser for the Treatment of Dermal or Mixed Type Melasma

DETAILED DESCRIPTION:
Primary Objective:

* To compare clinical efficacy by Modified MASI score between Fractional Picosecond 1,064 nm laser and daily application of 4% hydroquinone with 4% hydroquinone alone Secondary objectives
* To compare the clinical endpoints of Mexameter Melanin Index, brownish spot and Ultraviolet spots by VISIATM complexion analysis, The Antera 3D® imaging technology for pigmentation, quality of life by Dermatology Life Quality Index and patient's satisfaction between Fractional Picosecond 1,064 nm laser and 4% hydroquinone with 4% hydroquinone alone

ELIGIBILITY:
Inclusion Criteria:

* Female with melasma lesion on bilateral sides
* Age between 18-65 years
* Dermal or mixed type melasma, confirming by Wood's lamp test
* Willing to participant in this study and signed in informed consent form

Exclusion Criteria:

* Pregnancy / lactation
* Having an activity or working outside the building or unable to avoid heavy UV light
* Allergic to UV sunscreen, topical anesthetics , topical corticosteroid or hydroquinone Treatment with laser or chemical peeling within 3 months
* Treatment with Skin Lighting medication / food supplements within 4 weeks
* Currently use of topical retinoid, hydroquinone or corticosteroid within 4 weeks
* Use of whitening cream such as alpha arbutin, azelaic acid, kojic acid ascorbic acid or any cosmetics within 2 weeks
* Uncontrolled medical illness include non-skin cancers, coagulopathy
* Intra-cardiac device - pacemaker
* Photosentive conditions such as diabetes, thyroid disease, liver and kidney disease and photosensitive dermatosis
* Currently taking anticoagulant such as warfarin
* Active skin infection or acute dermatitis at testes skin sites
* Unable to follow and comply to the study protocol

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 30 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Modified MASI score | The mean change from the baseline to week-12 visit
Proportion of subjects with at least 50% MASI score improvement | from baseline to 12-week visit

SECONDARY OUTCOMES:
Mexameter Melanin index | baseline, week 4, week 8 and week 12
Global satisfaction score by Quartile rating scale | week 4, week 8 and week 12
Quality of life by DLQI | at week 12

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ho C, Nguyen Q, Lowe NJ, Griffin ME, Lask G. Laser resurfacing in pigmented skin. Dermatol Surg. 1995 Dec;21(12):1035-7. doi: 10.1111/j.1524-4725.1995.tb00554.x. PMID 7496671
- [Background] Weiss M, Weiss R, Lorden F, Trageser M, Beasley K. Picosecond laser for reduction of wrinkles: Long term results. Lasers Surg Med 2015; 47(S26): 24 (Abstract #68).